CLINICAL TRIAL: NCT03431909
Title: Evaluation Of Human Urinary Kallidinogenase in Acute Stroke Patients: Magnetic Resonance Spectrum and CT Perfusion
Brief Title: Evaluation Of HUK in Acute Stroke Patients: MRS and CTP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mrsctpzyf
Record Dates: First submitted 2017-12-05; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Human Urinary Kallidinogenase; Acute ischemic stroke; Magnetic resonance spectroscopy; CT perfusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kallikrein group (Experimental): Subjects receive kailikang treatment according to real clinical practice (suggest above 14 days treatment),0.15 peptide nucleic acids(PNA), once a day.
  Interventions: Drug: Human urinary kallidinogenase (HUK)
- Control group (Sham Comparator): Patients in control group will receive foundation treatment, including aspirin® (100 mg/d), clopidogrel® (75 mg/d), and atorvastatin® (20 mg/d) for 14 days
  Interventions: Drug: aspirin® , clopidogrel® , atorvastatin®

INTERVENTIONS:
Drug: Human urinary kallidinogenase (HUK) — Human urinary kallidinogenase can transform kininogen to bradykinin (kinin) and vasodilatory factors (kallidin)
  Arms: Kallikrein group
Drug: aspirin® , clopidogrel® , atorvastatin® — Patients in control group will receive foundation treatment, including aspirin® (100 mg/d), clopidogrel® (75 mg/d), and atorvastatin® (20 mg/d) for 14 days
  Arms: Control group

SUMMARY:
Background: Acute ischemic stroke (AIS) is a leading cause of morbidity and mortality worldwide. Human urinary kallidinogenase (HUK), a glycoprotein extracted from male urine currently used in China for enhancing cerebral perfusion5, plays a neuroprotective role including promoting angiogenesis, enhancing cerebral perfusion and suppressing the inflammatory response in animals and in patients with respect to regulating the kallikrein-kinin system. In previous clinical research, neurological function scores and cerebral perfusion scans were largely used to evaluate the efficiency of HUK. However, the mechanisms of Further well-conducted, randomized controlled studies using HUK are currently lacking.

Objective: To assess the Human urinary kallidinogenase effects on brain metabolite and cerebral perfusion changes using magnetic resonance spectroscopy and CT perfusion in patients with AIS.

Methods: The investigators plan to do a single-centre randomized, double-blind, controlled trial in which ischemic stroke patients will be randomized to treatment with either HUK or regular treatment within 72 hours of symptom onset. The study includes two MRS and two CTP scannings (before and after 2 week treatment) for all randomized subjects.

The endpoints will include improvement of the NIH Stroke Scale (NIHSS) score from baseline, modified Rankin scale (mRS) score and Barthel index at 14 days.

EvHUKMRS will test the following hypotheses:

1. HUK enhanced N-acetylaspartate (NAA) and cerebral blood flow (CBF) 14 days after treatment compared with control group.
2. HUK group compared to control group when administered 72 hours after onset of AIS improves recovery and functional outcome as assessed by improvement of NIHSS score , mRS score and BI score on day 14 post-stroke.

A positive result will have a significant impact in the management of AIS and pave the way for future studies aimed at finding the optimal dose and formulation of HUK for treating acute ischemic stroke.

DETAILED DESCRIPTION:
A)Specific Primary Objective:

1. To determine if HUK, administered within 72 hours of AIS onset is superior to regular treatment in improving NAA values and CBF on day 14 post stroke.

B) Specific Secondary Objectives:

1. To determine if HUK, administered within 72 hours of AIS onset is superior to regular treatment in reducing neurological deficit and improving functional outcome on day 14 post stroke.

Recruitment of study subjects:

Acute ischemic stroke patients admitted to the Neurology department in XWh (Xuan hospital) during the study period who are eligible to participate in this study based on criteria stated above will be invited to participate in this study.

The time window for enrolment will be within 72 hours of symptom onset. All eligible patients will be identified by the ward and on-call Neurology/Medical teams and referred to the study research assistants or investigators; who will then screen the patient for participation in this trial.

STUDY INTERVENTION The assigned treatment 0.15 PNA units of HUK injection or regular treatment will be administered once daily for 14 consecutive days soon after informed consent is taken and the patient is enrolled into the study.

Follow-up Assessment:

The neurologic deficits, global functional abilities and level of handicap will be scored using the NIH Stroke Scale (NIHSS) and the modified Rankin scale (mRS) at baseline and on day 14(plus or minus 14 days).

ELIGIBILITY:
Inclusion Criteria:

* ages ranging from 18 to 80 years
* onset time less than 72 h, NIHSS score ≥4;

Exclusion Criteria:

* TIA
* patients with contraindication of venous thrombolysis
* patients with encephalic bleeding disorder
* patients with incomplete hepatic and renal function
* patients with a medical history of peptic ulcer, haemorrhagic stroke, brain tumour or brain trauma
* patients who could not coordinate with an MRS scan and
* patients with vertebral basilar artery system infarction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
N-acetylaspartate as measured on Magnetic Resonance Spectrum study on admission | 14 days
  NAA Admit
Creatine as measured on Magnetic Resonance Spectrum study on admission | 14 days
  Cr Admit
Cholineas measured on Magnetic Resonance Spectrum study on admission | 14 days
  Cho

SECONDARY OUTCOMES:
The proportion of mordified Rankin Scale | 14 days
The proportion of NIHSS | 14 days
The proportion of mRS | 14 days
Cerebral blood flow as measured on CT perfusion study on admission | 14 days
  CBF Admit
Cerebral blood volume as measured on CT perfusion study on admission | 14 days
  CBV Admit
Mean transit time as measured on CT perfusion study on admission | 14 days
  MTT Admit
Time to peak as measured on CT perfusion study on admission | 14 days
  TTP Admit

CONTACTS AND LOCATIONS:
Overall Officials: Moli Wang, 1, Study Chair — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No